CLINICAL TRIAL: NCT01301222
Title: Randomized Controlled Trial on Role of Octreotide in Preventing Pancreatic Fistula and Complications After Pancreaticoduodenectomy in Patients With Soft Pancreas
Brief Title: Role of Octreotide in Preventing Pancreatic Fistula After Pancreaticoduodenectomy (PD) in Patients With Soft Pancreas
Acronym: PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PVS Memorial Hospital (Other)
Responsible Party: Principal Investigator, Dr Prakash K, Chief GI Surgeon, PVS Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVSMHEC
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Pancreatic Fistula
Keywords: octreotide; pancreatic fistula; soft pancreas; pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- octreotide (Experimental): octreotide arm 100mcg for 5 days. control has no octreotide
  Interventions: Drug: Inj. Octreotide

INTERVENTIONS:
Drug: Inj. Octreotide — 100 mcg subcutaneously for 5 days
  Other Names: Inj Octride

SUMMARY:
This randomized controlled trial (RCT) aims at assessing the influence of octreotide on pancreatic fistula or complications following pancreatoduodenectomy in patients with soft pancreas. Previously reported trials have included all types of pancreatic resections and have include all types of pancreas and have shown no clearcut benefit of octreotide after pancreaticoduodenectomy (PD). Soft pancreas and normal sized duct are the risk factors for fistula following PD. This study's focus is on this select group of patients and aims to assess the role of octreotide in patients with soft pancreas.

DETAILED DESCRIPTION:
Study design: Prospective open labeled randomized trial. AIM: Study aims at assessing the influence of octreotide on pancreatic fistula or complications following pancreatoduodenectomy in patients with soft pancreas.

ELIGIBILITY:
Inclusion Criteria:elective surgery patients undergoing pancreatoduodenectomy

* soft pancreas, no dilated duct

Exclusion Criteria:

* age > 75 years old
* documented chronic pancreatitis
* previous pancreatic surgery
* previous gastric surgery vagotomy
* documented pancreatic duct dilatation

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pancreatic fistula | 30 days
  All grades of postoperative pancreatic fistula as per ISGPF definition

SECONDARY OUTCOMES:
complications | 30 days
  All outcome measures like oral liquid feeds, semisolid food,hospital stay and complications like bleeding, intra-abdominal collections, respiratory complications, DGE etc are monitored

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Kurumboor, MS,MCh, Principal Investigator — GI Surgeon,PVS Memorial Hospital,Kochi, Kerala,India
Locations (1):
- PVS Memorial Hospital, Kochi, Kerala, India

REFERENCES:
- [Background] Vanounou T, Pratt WB, Callery MP, Vollmer CM Jr. Selective administration of prophylactic octreotide during pancreaticoduodenectomy: a clinical and cost-benefit analysis in low- and high-risk glands. J Am Coll Surg. 2007 Oct;205(4):546-57. doi: 10.1016/j.jamcollsurg.2007.05.011. Epub 2007 Aug 23. PMID 17903728
- [Background] Yeo CJ, Cameron JL, Lillemoe KD, Sauter PK, Coleman J, Sohn TA, Campbell KA, Choti MA. Does prophylactic octreotide decrease the rates of pancreatic fistula and other complications after pancreaticoduodenectomy? Results of a prospective randomized placebo-controlled trial. Ann Surg. 2000 Sep;232(3):419-29. doi: 10.1097/00000658-200009000-00014. PMID 10973392
- [Background] Suc B, Msika S, Piccinini M, Fourtanier G, Hay JM, Flamant Y, Fingerhut A, Fagniez PL, Chipponi J; French Associations for Surgical Research. Octreotide in the prevention of intra-abdominal complications following elective pancreatic resection: a prospective, multicenter randomized controlled trial. Arch Surg. 2004 Mar;139(3):288-94; discussion 295. doi: 10.1001/archsurg.139.3.288. PMID 15006886
- [Derived] Kurumboor P, Palaniswami KN, Pramil K, George D, Ponnambathayil S, Varma D, Aikot S. Octreotide Does Not Prevent Pancreatic Fistula Following Pancreatoduodenectomy in Patients with Soft Pancreas and Non-dilated Duct: A Prospective Randomized Controlled Trial. J Gastrointest Surg. 2015 Nov;19(11):2038-44. doi: 10.1007/s11605-015-2925-x. Epub 2015 Aug 25. PMID 26302879